CLINICAL TRIAL: NCT06502158
Title: Mifepristone Versus Misoprostol for Cervical Preparation Prior to Procedural Abortion at 12 to 16 Weeks' Gestation in an Academic Medical Center: a Randomized Controlled Pilot Trial
Brief Title: Mifepristone vs Misoprostol
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-15999
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Cervical Preparation
Keywords: Procedural Abortion; Surgical Abortion; Abortion, First Trimester; Cervical Dilators
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mifepristone (Experimental): Patients will be randomized to Mifepristone-alone in a 1:1 manner prior to procedural abortions. A paracervical block of 20 cubic centimeters (cc) 1% lidocaine, with or without vasopressin, will be administered in accordance with standard practices.
  Interventions: Drug: Mifepristone
- Misoprostol (Experimental): Patients will be randomized to Misoprostol-alone in a 1:1 ratio prior to procedural abortions. A paracervical block of 20cc 1% lidocaine, with or without vasopressin, will be administered in accordance with standard practices.
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Mifepristone — 200 milligrams (mg)
  Arms: Mifepristone
Drug: Misoprostol — 600 micrograms (ug)
  Other Names: Cytotec
  Arms: Misoprostol

SUMMARY:
The Investigator team hypothesizes that in a randomized trial comparing mifepristone-alone or misoprostol-alone for cervical preparation for procedural abortions at 12 to 16 weeks in hospital-based care, the proportion of patients who achieve successful cervical dilation will be different between the study groups.

DETAILED DESCRIPTION:
Cervical preparation is a critical component for the provision of safe abortion care in the later first trimester and beyond. The risk of surgical complications increases at 12 to 13 weeks gestation and routine use of cervical preparation is recommended. Cervical preparation options include misoprostol, mifepristone, and cervical dilators. Regimen choice is often guided by provider comfort, preference, or institutional guidelines. Misoprostol offers the advantage of facilitating same-day procedures, but side effects like pain and gastrointestinal symptoms can negatively affect patients' experiences. Furthermore, using misoprostol can pose logistical challenges in hospital-based main operating room environments, where abortions occur concurrently with all other surgical cases. Mifepristone is better tolerated than misoprostol but requires a multiple-day protocol for administration, which can pose logistical challenges.

Several studies demonstrate mifepristone's efficacy and safety as a cervical ripening agent for up to 16 weeks' gestation, however, despite its effectiveness, mifepristone for cervical preparation before procedural abortion has previously been limited by availability and cost. Recent studies demonstrating mifepristone's adjunctive benefit with osmotic dilators later in pregnancy, however, have broadened its use.

While most abortion care in the United States occurs in outpatient settings, about 3% occur in hospitals. This is expected to increase as the Dobbs versus Jackson Women's Health Organization decision exacerbates disparities in abortion access. In hospital-based abortion care, particularly at academic centers providing abortion training, there is a pressing need for innovative measures for cervical ripening. The Complex Family Planning Fellowship-trained faculty members at Montefiore will serve as research study surgeons. Cases will be performed in the main operating room under sedation or general anesthesia as determined by the anesthesiologist. A paracervical block of 20cc 1% lidocaine, with or without vasopressin, will be administered in accordance with standard practices.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish-speaking
* Capacity to consent
* Seeking induced abortion of a singleton pregnancy
* Between 12 weeks, 0 days and 16 weeks, 6 days (based on age at day of surgery)

Exclusion Criteria:

* History of more than two prior Cesarean deliveries
* Sonographic evidence of placenta previa
* Sonographic concern for morbidly adherent placenta
* Prior obstetric hemorrhage requiring transfusion
* Obstructive cervical or lower uterine segment fibroid
* Current therapeutic anticoagulation use
* Cerclage in situ
* History of more than one prior cervical excisional procedure
* BMI greater than 50 kg/m^2

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving Intended dilation | At time of surgery
  The proportion of participants achieving intended dilation at the start of the procedure will be summarized by treatment group and reported in percentages. Achievement of intended dilation will be determined by the attending surgeon. Overdilation resulting in passage of products of conception prior to time of surgery will be characterized as a treatment failure.

SECONDARY OUTCOMES:
Cervical dilation at start of procedure | Start of the Procedure
  Cervical dilation in centimeters (cm) at start of procedure will be summarized and reported using basic descriptive statistics.
Surgical time | Start to end of procedure, up to 4 hours
  Total surgical time will quantified and reported by treatment arm using basic descriptive statistics.
Estimated blood loss | Start to end of procedure, up to 4 hours
  Estimated blood loss will be quantified and reported per treatment arm using basic descriptive statistics.
Presence of Intraoperative Complications | From preoperative visit to discharge, up to 2 days
  The presence of peri-operative complications, defined as instances of hemorrhage, use of uterotonic medications, passage of products of conception prior to time of surgery, instances of extramural delivery, or need for unscheduled procedures, will be summarized and reported as "Yes" or "No" using basic descriptive statistics.
Patient Satisfaction | From preoperative visit to discharge, up to 2 days
  Patient Satisfaction will be assessed by responses to a survey administered in the Postoperative Care Unit (PACU) following the procedure. The patient will be asked to rate their satisfaction with the procedure on a 6-point Likert scale ranging from 0 (Not at all satisfied) to 5 (Most satisfied). Responses will be summarized by treatment group using basic descriptive statistics. Increased scores are associated with increased satisfaction.
Provider Satisfaction | From preoperative visit to discharge, up to 2 days
  Provider Satisfaction will be assessed by responses to a survey administered following the procedure. The care provider will be asked to rate their satisfaction with the procedure on a 6-point Likert scale ranging from 0 (Not at all satisfied) to 5 (Most satisfied). Responses will be summarized by treatment group using basic descriptive statistics. Increased scores are associated with increased satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Danvers, MD, MSCR, MBA, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allen RH, Goldberg AB. Cervical dilation before first-trimester surgical abortion (<14 weeks' gestation). Contraception. 2016 Apr;93(4):277-291. doi: 10.1016/j.contraception.2015.12.001. Epub 2015 Dec 9. PMID 26683499
- [Background] Kapp N, Lohr PA, Ngo TD, Hayes JL. Cervical preparation for first trimester surgical abortion. Cochrane Database Syst Rev. 2010 Feb 17;2010(2):CD007207. doi: 10.1002/14651858.CD007207.pub2. PMID 20166091
- [Background] Fox MC, Krajewski CM. Cervical preparation for second-trimester surgical abortion prior to 20 weeks' gestation: SFP Guideline #2013-4. Contraception. 2014 Feb;89(2):75-84. doi: 10.1016/j.contraception.2013.11.001. Epub 2013 Nov 11. PMID 24331860
- [Background] Ashok PW, Flett GM, Templeton A. Mifepristone versus vaginally administered misoprostol for cervical priming before first-trimester termination of pregnancy: a randomized, controlled study. Am J Obstet Gynecol. 2000 Oct;183(4):998-1002. doi: 10.1067/mob.2000.106767. PMID 11035353
- [Background] Borgatta L, Roncari D, Sonalkar S, Mark A, Hou MY, Finneseth M, Vragovic O. Mifepristone vs. osmotic dilator insertion for cervical preparation prior to surgical abortion at 14-16 weeks: a randomized trial. Contraception. 2012 Nov;86(5):567-71. doi: 10.1016/j.contraception.2012.05.002. Epub 2012 Jun 6. PMID 22682721
- [Background] Ohannessian A, Baumstarck K, Maruani J, Cohen-Solal E, Auquier P, Agostini A. Mifepristone and misoprostol for cervical ripening in surgical abortion between 12 and 14 weeks of gestation: a randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2016 Jun;201:151-5. doi: 10.1016/j.ejogrb.2016.04.007. Epub 2016 Apr 11. PMID 27132200
- [Background] Diedrich JT, Drey EA, Newmann SJ. Society of Family Planning clinical recommendations: Cervical preparation for dilation and evacuation at 20-24 weeks' gestation. Contraception. 2020 May;101(5):286-292. doi: 10.1016/j.contraception.2020.01.002. Epub 2020 Jan 31. PMID 32007418
- [Background] Ranji, U., Diep, K., & Salganicoff, A. (2023). Key Facts on Abortion in the United States. Retrieved from https://www.kff.org/womens-health-policy/report/key-factson- abortion-in-the-united-states/#Where-do-people-get-abortion-care.
- [Background] Jones RK, Kirstein M, Philbin J. Abortion incidence and service availability in the United States, 2020. Perspect Sex Reprod Health. 2022 Dec;54(4):128-141. doi: 10.1363/psrh.12215. Epub 2022 Nov 20. PMID 36404279